CLINICAL TRIAL: NCT05851235
Title: Results of a Programme of Intensive Prehabilitation in GEriatric Patients Operated for Colo-Rectal Neoplasia
Brief Title: Prehabilitation in Geriatric Patients With Colorectal Neoplasia
Acronym: PIGEON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Istituto Oncologico Romagnolo (IOR) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRST153.08
Record Dates: First submitted 2023-03-22; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-03

CONDITIONS: Colo-rectal Cancer
Keywords: Prehabilitation
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal cancer patients (Experimental): Patients with colon or rectal cancer awaiting surgery
  Interventions: Other: Prehabilitation course

INTERVENTIONS:
Other: Prehabilitation course — During prehabilitation course, patients will follow a nutritional programme, a cardiovascular and motor programme and a psychological programme.

SUMMARY:
This an interventional, non-pharmacologic study. Prehabilitation is a multidisciplinary preoperative intervention aimed at preventing or reducing functional decline related to surgery and improving perioperative outcomes. The current study is aimed at standardizing a prehabilitation pathway, evaluating its feasibility within the AUSL Romagna in collaboration with the PRIME Centre and the multiple professions that populate the two institutes in the spirit of confirming the beneficial effect of an integrated prehabilitation programme on surgical outcomes.

Patients will follow an intensive prehabilitation course before surgery:

* Colon cancer patients will do 4 weeks of prehabilitation before surgery.
* Rectal cancer patients will do 12 weeks of prehabilitation after neoadjuvant therapy and before surgery.

The prehabilitation course is structured around the following aspects:

* Frailty assessment and identification of optimisation fields
* Optimisation of modifiable factors (anaemia, polypharmacotherapy, smoking, alcoholism, diabetes)
* Assessment by an integrative medicine specialist
* Nutritional pre-qualification
* Cardiovascular, respiratory, motor prehabilitation
* Emotional and psychological prehabilitation

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
2. Male/female participants who are at least 70 years of age on the day of signing informed consent.
3. Patients with confirmed diagnosis of colorectal cancer awaiting major surgery.

Exclusion Criteria:

1. Clinical need for emergency intervention.
2. Severe cognitive impairment (MMSE<20*)
3. Severe dependency (ADL<3)
4. Stage IV colorectal neoplasia

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible participants completed the personalized proposed prehabilitation program | 4 months
  The primary endpoint of the study will be the feasibility of delivering a prehabilitation program, based on adherence. This study will be deemed as feasible if ≥80% of eligible participants completed the personalized proposed prehabilitation program.

SECONDARY OUTCOMES:
Adherence to prescription | 4 months
  Percentage of patients with compliance greater than 80% to prehabilitation prescription
30-days mortality | 30 days after the surgery
  Proportion of patients who died for all causes within 30 days after the surgery
Overall morbidity rate and major morbidity rate | 4 months
  Calculated according Clavien-Dindo classification
Preservation/improvement of pre-operative quality of life before vs. 1-month after surgery | 30 days after the surgery
  Questionnaire EQ-5D-3L. Test results are presented in the form of an index and a VAS scale. The index is based on patients' quality of life in 5 domains across 3 levels. Distribution of EQ-5D-3L dimension responses at different times were calculated. The index, which is a value attached to an EQ-5D-3L profile according to a set of weights that reflect, on average, people's preferences about how good or bad the state is, ranges from 0 (poorest quality of life) to 1 (perfect health). The value set generated from the European population (EQ) was used as the reference cohort for index calculation.
  The VAS score is generated by asking the patient how he/she ranked his/her QoL, as compared to his/her peers, on a scale from 0 to 100, where higher values were associated to a better quality of life. EQ-5D-3L index and VAS were expressed as mean (Standard Deviation-SD) and median (minimum-maximum), while frequency will be calculated for categorical variables (five domains of EQ-5D-3L).
Preservation/improvement of pre-operative quality of life before vs. 1-month after surgery. | 30 days after the surgery
  Questionnaire EORTC QLQ-ELD14, a questionnaire that comprise five scales (mobility, worries about others, future worries, maintaining purpose and burden of illness) and two single items (joint stiffness and family support). Four levels were available for the response (1=not at all, 2=a little, 3=quite a bit, 4=very much). Distribution of EORTC QLQ-ELD14 items at different times were calculated. All scale and item scores are transformed to a 0-100 scale, higher scores representing a worse outcome except for maintaining purpose and family support.
  EORTC QLQ-ELD14 scores were expressed as mean (Standard Deviation-SD) and median (minimum-maximum), while frequency will be calculated for categorical variables (for the five scales and two single items).
Postoperative functional recovery at one month after surgery | 30 days after the surgery
  Percentage of patients experiences functional recovery as described in protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Isacco Montroni, MD, Study Chair — AUSL della Romagna
Locations (1):
- AUSL della Romagna, Ravenna, RA, Italy